CLINICAL TRIAL: NCT06206629
Title: Evaluation of Contralateral R1 Component of the Blink Reflex in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Contralateral R1 in Amyotrophic Lateral Sclerosis
Acronym: MOTOBLINK
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1291
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; ALS; Electroneuromyography; ENMG
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALS patients: Patients with ALS (Awaji criteria)
  Interventions: Diagnostic Test: blink reflex evaluation
- Non-ALS patients: Patients referred to the neurophysiology unit for a suspicion of ALS du to motor weakness, but in whom the diagnosis is ruled out.
  Interventions: Diagnostic Test: blink reflex evaluation
- Healthy volunteers: Healthy volunteers who will undergo a blink reflex evaluation on ENMG.
  Interventions: Diagnostic Test: blink reflex evaluation

INTERVENTIONS:
Diagnostic Test: blink reflex evaluation — A blink reflex evaluation will be performed in all subjects

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease affecting both upper and lower motor neurons. Electroneuromyography is an important tool for the diagnosis. Previous studies have shown that different components of the blink reflex, such as the latencies of homo- and contralateral R2 responses can be affected. Studies have found that a contralateral R1 component can appear in neurological diseases with affection of the central nervous system especially upper motor neuron, such as HTLV1 infection. Thus, you aim to determine if a contralateral R1 component could be present in ALS.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Aged 18 to 99 years old
* Referred for suspected motor neuromuscular disease
* Collection of non-opposition

For healthy subjects:

* Aged 18 to 99 years old
* Absence of any neurological pathology
* Collection of non-opposition

Exclusion Criteria:

* Previous damage linked to another cause of the cranial nerves
* Prior brainstem lesions
* Persons deprived of liberty by a judicial or administrative decision
* Patient under judicial protection, unable to express consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the neurophysiology unit from the Hospices civils de Lyon, for a suspicion of motor neuron disease.
  And healthy volunteers for the third group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Presence of a contralateral R1 component on blink reflex evaluation. | Day 1
  A blink reflex evaluation will be performed in all subjects : Blink reflex will be recorded with surface electrodes placed medially over the lower part of the eyelid, on the orbicularis oculi muscle, with a reference electrode 2 cm laterally. Stimuli will be delivered to the supraorbital nerve by surface electrodes with an intensity required to generate a consistent homolateral R1 response.
  A contralateral R1 component will be defined as an early compound muscle action potential recorded in the contralateral orbicularis oculi muscle.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No